CLINICAL TRIAL: NCT04597931
Title: Evaluation of Romosozumab vs. Zoledronic Acid Effect in Patients With Spinal Cord Injury and Low Bone Mineral Density
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Liana Tripto Shkolnik, Deputy Director, Division of Endocrinology, Diabetes and Metabolism, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-20-7186-LT-CTIL
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Osteoporosis Fracture; Spinal Cord Injuries
Keywords: bone mineral density; fracture; romosozumab
MeSH Terms: conditions — Osteoporotic Fractures; Spinal Cord Injuries; Fractures, Bone | interventions — romosozumab; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC Romosozumab 210 mg/monthly (Experimental): SC Romosozumab 210 mg/monthly
  Interventions: Drug: Romosozumab
- IV Zoledronic acid 5 mg (Active Comparator): IV Zoledronic acid 5 mg
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Romosozumab — SC Romosozumab 210 mg/monthly
  Arms: SC Romosozumab 210 mg/monthly
Drug: Zoledronic Acid — IV Zoledronic acid 5 mg
  Arms: IV Zoledronic acid 5 mg

SUMMARY:
This is a randomized study to determine the effects of monthly romosozumab for one year or one-time zoledronic acid on bone mineral density (BMD) and biochemical markers of bone formation and resorption, in patients with spinal cord injury (SCI) and low BMD.

DETAILED DESCRIPTION:
This is a randomized open-label study to determine the effects of monthly romosozumab for 12 month or one-time zoledronic acid infusion on bone mineral density (BMD) and biochemical markers of bone formation and resorption, in patients with spinal cord injury (SCI) and low BMD.

Patients: Thirty women between 20-70 years of age with spinal cord injury and low bone mass (BMD T-score lower than -2.0 in at least one location: Lumbar Spine, Femoral Neck or Total Hip sites) will receive study medication.

Primary outcome:

Total hip BMD change during a one-year treatment period.

Secondary outcome:

Change in Femoral neck BMD at 12 months, Bone turnover markers change over time (3, 9 and 12 month): C-terminal telopeptide of type I collagen (CTX), N-terminal propeptide of type I procollagen (P1NP).

Study population:

Thirty women between 20-70 years of age with spinal cord injury that occurred more than 24 month ago and low bone mass (BMD T-score lower than -2.0 in at least one location: Lumbar Spine, Femoral Neck or Total Hip sites)

ELIGIBILITY:
Inclusion Criteria:

* BMD T-score ≤ -2.0 at the lumbar spine, total hip or femoral neck
* SCI of at least 24-month but less than 7 years duration,
* American Spinal Injury Association (ASIA) Impairment Scale A-C

Exclusion Criteria:

* myocardial infarction (MI) or stroke within the preceding year
* high cardiovascular risk, 10 years Framingham score over 20 %.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Total hip BMD change during a one-year treatment period | one year
  BMD change

SECONDARY OUTCOMES:
Change in Femoral neck BMD at 12 months | one year
  BTM change
Bone turnover markers change | one year
  Bone turnover markers change over time (3, 9 and 12 month)

CONTACTS AND LOCATIONS:
Overall Officials: Liana Tripto-Shkolnik, MD, Principal Investigator — Sheba Medical Center, Tel Hashomer

IPD SHARING:
Plan to Share IPD: No